CLINICAL TRIAL: NCT04625504
Title: Investigating Biological Targets, Markers, and Intervention for Chronic Pain
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Vanderbilt University Medical Center (Other)
Responsible Party: Principal Investigator, Poppy Schoenberg, Principle Investigator, Vanderbilt University Medical Center
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Basic Science
Other Study IDs: IRB #201646
Record Dates: First submitted 2020-10-29; First posted 2020-11-12 (Actual); Last update posted 2023-03-27 (Actual); Status verified 2023-03

CONDITIONS: Chronic Pain; Pain, Chronic; Pain Syndrome; Pain, Neuropathic; Pain, Intractable
Keywords: Neurophysiology; Endocrine; EEG/ERP; Cognitive; Mindfulness; Mechanistic Clinical Trial
MeSH Terms: conditions — Chronic Pain; Somatoform Disorders; Neuralgia; Pain, Intractable

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Mindfulness Based Intervention (MBI) (Experimental): Patients Active Intervention group
  Interventions: Behavioral: Mindfulness Based Intervention
- Wait-list Control (WL) (No Intervention): Patients Control receiving no treatment
- Healthy Control (HC) (No Intervention): Healthy Control receiving no treatment

INTERVENTIONS:
Behavioral: Mindfulness Based Intervention — Standardized 8-week Cognitive and Behavioral Psychotherapy group with 26 hrs of in-class training and homework, along with 1 all-day retreat in which core mindfulness skills are developed
  Other Names: MBI
  Arms: Mindfulness Based Intervention (MBI)

SUMMARY:
This multi-modal methods study will investigate neurophysiological, endocrinological, cognitive, psycho-social-emotional markers of chronic pain, and therapeutic targets using integrative health treatments.

DETAILED DESCRIPTION:
It is estimated that 50 million adults in the USA suffer from chronic pain. Chronic pain is one of the most common reasons adults seek medical care, causing undue burden on primary care channels and treatment costs. Chronic pain is associated with (1) restrictions in mobility and daily activity, (2) dependence on opioids, (3) anxiety and depression, and (4) poor perceived health and reduced quality of life. Developing robust and specific non-pharmacologic intervention programs, on par with pharmacological clinical outcomes without harmful side-effects, addictive risk, and toxicity, is a crucial unmet clinical need and a research priority for the NCCIH. Understanding the mechanistic pathways of these interventions is key to their clinical development and implementation for treating chronic pain in primary care.

Mindfulness-Based Interventions (MBIs) show similar clinical efficacy for mood disorders as pharmacology, and co-morbid symptoms of depression and anxiety. Meta-analysis including 183 patients with Multiple Sclerosis showed efficacy in psychosocial outcomes, quality of life, anxiety, depression, and select physical symptoms including fatigue, pain, and vestibular symptoms. The clinical efficacy of MBIs appears to extend mood disorders, as a systematic review including 13 studies in fibromyalgia, chronic fatigue, and irritable bowel syndrome showed significant effect sizes, reported as standardized mean difference (SMD), compared to control conditions in reducing symptom severity (SMD= -.40), and pain (SMD= -.21). Cognitively, MBIs appear to enhance executive control and self-regulatory processing, that has a beneficial effect upon emotion regulation, pain perception, and has shown to reduce ruminative ideation. Previous research has also suggested that mindfulness meditation training improves chronic pain symptomology through certain mechanisms such as disengagement from pain-related threats. While previous research has shown MBIs to be effective in treating certain health conditions, the mechanisms by which MBIs lead to clinical changes remain unclear. No study has adequately investigated biological or neurophysiological markers in chronic pain that may correlate with reduction in clinical symptoms.

This overarching study aims to identify key phenotypic markers and treatment targets of chronic pain, and further understand MBI mechanism in its treatment.

ELIGIBILITY:
Inclusion Criteria for Chronic Pain Patients:

* Age range: 18-60 years
* Must indicate pain intensity of 3/10 and must have experienced pain for at least 3 months
* Must possess English language skills sufficient for providing informed consent, completing questionnaires, and understanding instructions
* Must have a stable medication regimen or no medication or dosage changes within the past month

Blood Collection Inclusion:

* At least 110 pounds
* Generally healthy by self-report on day of collection (i.e., free of cold and flu symptoms on the day of collection, no infections within two weeks prior to collection, no known sickle cell disease)
* Including the study draw, blood donation for clinical or research purposes within the preceding eight weeks will not exceed 550 mL
* No more than one blood draw will have occurred during the preceding week

Exclusion Criteria for Chronic Pain Patients:

* Prior diagnosis of bipolar I, bipolar II, psychotic personality disorder, borderline personality disorder, and/or narcissistic personality disorder
* Current history (equal/less than 6 months) of substance abuse/dependence
* Current history (equal/less than 6 months) of regular meditation practice (>1 session/week; >10 min/session)
* Diagnosis of bipolar I, bipolar II, psychotic personality disorder, borderline personality disorder, and/or narcissistic personality disorder
* History of medical illness associated with possible changes in cerebral tissue or cerebrovasculature (e.g., stroke) or with neurologic abnormality (e.g., seizure disorder, cerebrovascular or neoplastic lesion, neurodegenerative disorder, or significant head trauma, defined by loss of consciousness of ≥ 5 minutes)
* Current suicidal ideation

Exclusion Criteria for Healthy Controls:

* Current history (equal/less than 6 months) of substance abuse/dependence
* No major medical illness. History of medical illness associated with possible changes in cerebral tissue or cerebrovasculature (e.g., stroke) or with neurologic abnormality (e.g., seizure disorder, cerebrovascular or neoplastic lesion, neurodegenerative disorder, or significant head trauma, defined by loss of consciousness of ≥ 5 minutes)
* Current suicidal ideation
* Current history (equal/less than 6 months) of regular meditation practice (>1 session/week; >10 min/session)

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 69 (Actual)
Dates: Start 2020-11-25 (Actual); Primary Completion 2022-07-28 (Actual); Study Completion 2022-07-28 (Actual)

PRIMARY OUTCOMES:
Electroencephalography (EEG) | 36 months
  Oscillatory Activity
Electroencephalography (EEG) | 36 months
  Event-Related Potentials (ERPs)

SECONDARY OUTCOMES:
Endocrine Measures | 36 months
  Cortisol, Oxytocin
Cognitive-Behavioral Measure | 36 months
  Executive Inhibitory Control
Cognitive-Behavioral Measure | 36 months
  Working Memory

OTHER OUTCOMES:
Clinical: Pain Measure | 36 months
  McGill Pain Questionnaire; Score range: 0 -- 45, with higher scores indicating worse outcomes.
Clinical: General Symptoms | 36 months
  Patient Reported Outcomes Measurement Information System; Score range: 4 -- 20, with higher scores indicating worse outcomes
Clinical: Mindfulness Skills | 36 months
  Five Facet Mindfulness Questionnaire; 5 domains, Score range: 0 -- 8, with higher scores indicating more mindfulness skills.
Clinical: Interoception | 36 months
  Multidimensional Assessment of Interoceptive Awareness; 8 subdomains, Score range: 0 -- 5, with higher scores indicating more interoceptiveness

CONTACTS AND LOCATIONS:
Overall Officials: Poppy LA Schoenberg, PhD, Principal Investigator — Vanderbilt University Medical Center
Locations (1):
- Vanderbilt University Medical Center, Nashville, Tennessee, United States

IPD SHARING:
Plan to Share IPD: Yes
The PI will adhere to the NIH Sharing of Biomedical Research Resources: Guidelines for Recipients of NIH Grants and Contracts on Obtaining and Disseminating Biomedical Research Resources.
  1. Quality-controlled raw data as well as processed data used in publications will be de-identified before sharing upon "reasonable request". As described in the proposal, workflows and structure will be exactly described in reports and documented to allow precisely reproduce results from raw data and replicate methodology. Final data (computerized datasets with raw data and derived variables) that have not yet been published will be shared in a timely manner.
  2. Software programs (i.e. experimental paradigm scripts produced for this study) and documentation will be made available for research purposes to replicate findings upon "reasonable request", and any software/script sharing requirements by journals.
Supporting Information: CSR
Time Frame: 48 months